CLINICAL TRIAL: NCT05847595
Title: Implicit Versus Explicit Motor Training for Upper Extremity Rehabilitation in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Anwar (Other)
Responsible Party: Sponsor-Investigator, Ahmed Anwar, Assistant Lecturer of physical Therapy, Egyptian Chinese University (ECU), Egyptian Chinese University
Organization: Egyptian Chinese University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004192
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: CVA (Cerebrovascular Accident)
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group A (Sham Comparator): will be treated by selected physical therapy program only for 60 minutes.
  Interventions: Other: Selected physical therapy program
- Study group B (Experimental): will be treated by implicit motor training program for 30 minutes, in addition to the conventional physical therapy program for the lower extremity for 30 minutes ,total duration 60 minutes.
  Interventions: Other: Implicit motor training program; Other: Selected physical therapy program
- Study group C (Experimental): will be treated by explicit motor training program for 30 minutes, in addition to the conventional physical therapy program for the lower extremity for 30 minutes, total duration 60 minutes.
  Interventions: Other: Explicit motor training program; Other: Selected physical therapy program

INTERVENTIONS:
Other: Implicit motor training program — The implicit motor training aims to create a learning situation in which the learner is not (or minimally) aware of the underlying rules of the practiced motor skill. Cognitive-motor dual-task training will be used, which involves practicing hand-reaching and grasping in different locations in space while performing cognitive tasks associated with attention, memory, and executive function. The cognitive tasks include naming words, counting backwards, counting tones, counting days and months backwards, listening to a number and counting backwards by twos and threes, telling daily stories, spelling words backward, continuous subtraction of 7 from 100, and the Stroop task. The training will be tailored to the participant's abilities.
  Arms: Study group B
Other: Explicit motor training program — The explicit motor training aims to create a learning situation in which the learner is very aware of the learning process by providing detailed explicit instructions on each exercise. The Motion Guidance Shoulder Kit will be used for this intervention, which involves four exercises: "Around the clock" in flexion and abduction, "Locate the Target" in active range of motion, "Butterfly" in tracing small and large butterfly patterns, and "Test your positional awareness" in locating circles with eyes open and closed. The kit involves a strap around the forearm with a laser to guide the movement of the arm during the exercises.
  Arms: Study group C
Other: Selected physical therapy program — The selected physical therapy program, which includes shoulder joint mobilization, graduated active exercises for shoulder muscles, hand weight bearing exercises, Approximation of the upper limb joints. While, the conventional physical therapy program for the lower extremity which includes gait training, strengthening exercises and balance training .

SUMMARY:
Training methods that improve proprioception of the shoulder joint involve specific tasks targeting joint position sense, kinesthesia, or sense of force. These exercises can involve explicit or implicit motor learning. Explicit learning involves verbal knowledge of movement performance, while implicit learning involves minimal verbal knowledge and learning in a less conscious manner. The purpose of the study is to identify the efficacy and difference between implicit and explicit motor training in improving upper extremity functions in chronic stroke patients. The study will use laser pointer pattern tracking exercises and precise repositioning tasks for explicit motor training and a cognitive-motor dual-task training for implicit motor training. The laser-pointer assisted angle reproduction test, Wolf Motor Function Test and Arm Motor Ability Test will be used for evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Age is ranging between 50 to 65 years
2. Diagnosis of a single stroke 6 months to 2 years prior to study entry confirmed by neuroimaging reports (to minimize the chance that improvements occur because of spontaneous recovery).
3. Sufficient cognitive and language abilities to understand and follow multiple-step instructions (a score of 24 or more on the mini mental state examination).
4. Adequate vision to track the laser beam.
5. Muscle strength of ≥ 3/5 for all upper extremity joints on manual muscle testing.
6. Subjects are able at least to partially move outside of synergies at the affected elbow (Brunnstrom recovery stage in the upper limb following stroke is 4 or greater)
7. Spasticity at the paretic elbow, wrist, or fingers, defined as a score less than 2 on the modified Ashworth scale.

Exclusion Criteria:

1. Uncontrolled seizure disorders.
2. Additional neurological impairments, for example, Parkinson disease that (severely) influence their upper limb functions.
3. Excessive spasticity at the paretic upper limb muscles defined as a score equal or more than 2 on the modified Ashworth scale.
4. Excessive pain in the affected UE, as measured by a score of 5 or higher on a 10-point visual analog scale.
5. Patients with musculoskeletal disorders of upper limb joints, such as severe arthritis, fractures, or fixed deformities.
6. Patients with cognitive, visual, or auditory impairments.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Upper extremity motor ability | 4-weeks
  Wolf Motor Function Test
ADL functions of the upper extremity | 4-weeks
  Arm Motor Ability Test

SECONDARY OUTCOMES:
Shoulder joint proprioception | 4-weeks
  laser-pointer assisted angle reproduction test

CONTACTS AND LOCATIONS:
Locations (1):
- Egyptians Chinese University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided